CLINICAL TRIAL: NCT06593431
Title: Extending Outcomes for Pancreas Cancer Patients With Nominal Oligometastatic Disease (EXPAND): A Randomized Phase III Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1159; NCI-2024-07461 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-08-31; First posted 2024-09-19 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Pancreas Cancer; Oligometastatic
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MDT (Metastasis-Directed Therapy) (Experimental): Patients will be randomized 1:1 to (a) MDT or (b) systemic therapy alone (no MDT).
  Interventions: Radiation: Consolidative Radiation
- System Therapy (control) (Experimental): Patients will be randomized 1:1 to (a) MDT or (b) systemic therapy alone (no MDT).
  Interventions: Radiation: Consolidative Radiation

INTERVENTIONS:
Radiation: Consolidative Radiation — Participants will receive treatment through radiation therapy

SUMMARY:
The EXPAND trial (EXtending outcomes for PAncreas cancer patients with Nominal oligometastatic Disease) is a randomized phase III trial assessing the efficacy of MDT to improve PFS and OS for patients with oligometastatic pancreatic ductal adenocarcinoma (PDAC).

DETAILED DESCRIPTION:
Primary Objectives:

To determine whether, in patients with oligometastatic pancreatic ductal adenocarcinoma, MDT to all sites of disease confers a benefit in PFS compared to systemic therapy alone.

Secondary Objectives:

Key secondary objective: To determine whether, in patients with oligometastatic pancreatic ductal adenocarcinoma, MDT to all sites of disease confers a benefit in OS compared to systemic therapy alone.

To assess safety/tolerability of MDT in patients with oligometastatic PDAC.

To assess time to new lesion formation between treatment arms.

To assess time to next-line systemic therapy between treatment arms.

To assess incidence and duration of time off systemic therapy between treatment arms.

To assess incidence and duration of time on maintenance systemic therapy between treatment arms.

To assess time to local failure between treatment arms for lesions present at enrollment/baseline.

To compare quality of life (QOL) between treatment arms.

To assess the above primary and secondary objectives, as well as exploratory objectives, which may be differential based on receipt of different forms of MDT in the MDT arm (e.g,. surgery, external beam radiotherapy, etc).

Exploratory Objectives:

To identify predictive/prognostic biomarkers correlated with a benefit for MDT.

To investigate changes in biomarker profile over time and in response to MDT.

ELIGIBILITY:
Inclusion Criteria:

Age 18

Histologically or cytologically confirmed pancreatic ductal adenocarcinoma.

Histologic / cytologic confirmation of pancreatic ductal adenocarcinoma may come from the primary tumor (i.e., via FNA at initial diagnosis). Histological/pathologic confirmation of distant metastatic disease is not required if clinical and radiographic consensus is that the patient has distant metastatic disease.

Eastern Cooperative Oncology Group (ECOG) performance status ≤2

Candidate for MDT (including radiation therapy, surgical resection, ablation, and embolization) to all sites of disease including oligometastatic sites and if present intact primary / regional nodal disease.

Between one and five distant metastatic lesions, counted as follows: each lesion (not site) will be counted as one, with the exception of metastatic lymph node stations, which will collectively count as one lesion. Regional nodal stations will be counted as a collective single lesion if present. All progressive lesions must be amenable to local therapy as noted in criterion 4.2.1.4 above.

Counting of oligometastatic nodal disease will be based on nodal chains. A nodal chain will be considered a single metastatic lesion if the presence of that node results in the patient as having M1 disease per the TNM staging system, AJCC version 8.0. In addition, one of the following criteria must be met: a) ≥1 LN meets radiologic criteria for metastatic disease via RECIST 1.1 (short axis ≥15mm), b) pathologic assessment has confirmed the presence of metastatic cancer cells, and/or c) the LN exhibits imaging signal characteristic of a metastatic lesion (e.g. FDG avidity, contrast enhancement, etc.). In the event of ambiguity or equivocal findings, the principal investigator or co-principal investigator will make a final determination of whether criteria are met. The following caveats apply:

In patients with a LN exhibiting a short axis ≥15mm and who have other diagnoses that can produce enlarged LNs (e.g. indolent CLL, sarcoidosis, etc…) or a prior history of benign enlarged LNs will not be considered to have metastatic disease per the discretion of the treating physician.

LN chains that occur bilaterally will be considered separate metastatic sites. For example, left axilla LNs will counted separately from right axilla LNs.

The following midline LN chains will be counted as 1 metastatic site: mediastinal, para-aortic, mesenteric.

The following bilateral LN chains will be counted as 1 metastatic site for unilateral involvement, and 2 for bilateral for involvement: preauricular, cervical and occipital, supraclavicular, infraclavicular, pectoral, axillary, hilar, epitrochlear and brachial, iliac, inguinal and femoral, popliteal.

Baseline imaging must include a scan done within 4 weeks prior to randomization, demonstrating oligometastatic disease by RECIST (v1.1) criteria compared to pre-baseline imaging.

Baseline imaging must be done within 4 weeks prior to randomization, and the following imaging is required: PET/CT scan or CT scan of the chest/abdomen/pelvis. MRI may be substituted as indicated (i.e., CT scan of chest plus MRI abdomen/pelvis).

Diagnostic laparoscopy may be indicated prior to enrollment if any concern for peritoneal disease / carcinomatosis is present, at the investigator's discretion. Presence of peritoneal carcinomatosis will exclude the patient from this trial as below. Indications for peritoneal carcinomatosis may include findings concerning for but not definitive for peritoneal disease on diagnostic imaging, elevated CA-19-9, and clinical symptoms concerning for peritoneal disease.

Patients referred for the study that require immediate MDT can receive treatment to CNS lesions or other symptomatic lesions prior to randomization, but these lesions will be counted towards the total number of oligometastatic lesions.

Patients with >5 discrete metastatic sites previously with subsequent 'induction' of oligometastatic disease (<=5 discrete sites; induction via response to systemic therapy) may be eligible if 5 or fewer metastatic disease sites have been present / noted radiographically for a minimum of 6 months, and pending principal investigator review/discretion.

Females of childbearing potential must not be breast feeding and must have a negative serum or urine pregnancy test and must agree to use adequate contraception from the time of screening until 3 months after discontinuation of the study medication. Acceptable methods of contraception include total and true sexual abstinence, tubal ligation, hormonal contraceptives that are not prone to drug-drug interactions (IUS Levonorgestrel Intra Uterine System (Mirena), Medroxyprogesterone injections (Depo-Provera), copper-banded intra-uterine devices, and vasectomized partner. All hormonal methods of contraception should be used in combination with the use of a condom by their sexual male partner. Females of childbearing potential are defined as those who are not surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause). Women will be considered post-menopausal if they have been amenorrheic for the past 12 months without an alternative medical cause. The following age-specific requirements must also apply: Women < 50 years old: they would be considered post-menopausal if they have been amenorrheic for the past 12 months or more following cessation of exogenous hormonal treatments. The levels of Luteinizing Hormone (LH) and Follicle-Stimulating Hormone (FSH) must also be in the post-menopausal range (as per the institution). Women ≥ 50 years old: they would be consider post-menopausal if they have been amenorrheic for the past 12 months or more following cessation of all exogenous hormonal treatments, or have had radiation-induced oophorectomy with the last menses > 1 year ago, or have had chemotherapy-induced menopause with >1 year interval since last menses, or have had surgical sterilization by either bilateral oophorectomy or hysterectomy.

Non-sterilized males who are sexually active with a female partner of childbearing potential must use adequate contraception for the duration of the study and 6 months after the last dose of study medication. Adequate contraception methods include: birth control pills (e.g. combined oral contraceptive pill), barrier protection (e.g. condom plus spermicide, cervical/vault cap or intrauterine device), and abstinence. Patients should not father a child for 6 months after completion of the study medication. Patients should refrain from donating sperm from the start of dosing until 6 months after discontinuing the study medication. If male patients wish to father children they should be advised to arrange for freezing of sperm samples prior to the start of the study medication.

Demonstration of adequate organ function as defined in the table below, all screening labs to be performed within 4 weeks prior to study enrollment:

Exclusion Criteria

Metastatic effusion (e.g. pleural effusion or ascites). Note that patients with an effusion that is too small to sample will be eligible for the trial.

Leptomeningeal disease.

Peritoneal carcinomatosis.

Cognitively impaired subjects (e.g. inability to sign informed consent.)

Any condition that, in the opinion of the investigator, would interfere with the study treatment or interpretation of the study results.

Diffuse bone marrow involvement as defined by disease involvement of a BM biopsy from a site that does not have radiologic evidence of a bone metastasis.

More than 4 prior lines of systemic therapy to treat metastatic disease.

Diagnosis of active scleroderma, lupus, or other rheumatologic disease which in the opinion of the treating radiation oncologist precludes safe delivery of radiotherapy. Such patients may be eligible if dispositioned to non-radiotherapy MDT.

Known psychiatric or substance abuse disorder/s that would interfere with trial participation.

Concurrent (synchronous or metachronous) other primary malignancy that in the opinion of the treating physician team presents a substantial risk to the patient's life as a competing risk of death (against the primary oligometastatic pancreatic cancer being considered for MDT as part of this trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2029-06-29 (Estimated); Study Completion 2029-06-29 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Ludmir, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org